CLINICAL TRIAL: NCT00334269
Title: Study of Health Assessment and Risk Evaluation (SHARE) in Aboriginal Peoples (AP) Action Toward Obesity Prevention (SHARE-AP Action)
Brief Title: Study of Health Assessment and Risk Evaluation in Aboriginal Peoples Action Toward Obesity Prevention (SHARE-AP Action)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Population Health Research Institute (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MCT64076; ISRCTN86187625; CIHR Grant No. MCT64076; Final Protocol Nov.20, 2003
Record Dates: First submitted 2006-06-06; First posted 2006-06-07 (Estimated); Last update posted 2009-09-29 (Estimated); Status verified 2009-09

CONDITIONS: Obesity
Keywords: obesity; physical activity; daily energy intake; nutrition; healthy lifestyle; Aboriginal; body fat; exercise; education; family; body mass index; knowledge; randomized controlled trial; community; intervention; Six Nations Indian Reserve; household; health counselling
MeSH Terms: conditions — Obesity; Motor Activity | interventions — Nutritionists

INTERVENTIONS:
Behavioral: Health messaging at weekly home visits by health counsellor
Behavioral: Weekly home delivery of bottled spring water
Behavioral: Weekly afterschool physical activity program for 5-18y.o.
Behavioral: Cooking classes and grocery store tours with dietician
Behavioral: Pedometers to track/increase weekly physical activity

SUMMARY:
The purpose of this study is to develop an effective intervention strategy to prevent & reduce obesity among a high risk cohort of Aboriginal families.

DETAILED DESCRIPTION:
Obesity is a major public health problem in North America. The most recent estimates indicate that over 35% of men and 27% of women over the age of 18 are obese (body mass index (BMI) ≥30), and the prevalence of obesity among children and adolescents has increased over the last two decades to about 13%. Obesity leads to a number of chronic health problems including diabetes, hypertension, cardiovascular disease (CVD), and some cancers. Throughout the world, Aboriginal people suffer a high prevalence of overweight and obesity. This is likely due to their transition from a lifestyle of modest energy intake and high levels of physical activity, to a lifestyle of high energy intake and low levels of physical activity. This in turn has led to extraordinarily high rates of overweight, obesity, and type 2 diabetes.

There is an urgent need to test interventions to reduce or prevent obesity among Aboriginal people. Obesity has been resistant to traditional public health education strategies and novel approaches at multiple levels to develop effective strategies are required. SHARE-AP ACTION is a randomized controlled trial testing if a household-based intervention to improve change dietary and physical activity patterns has the potential to succeed where individual, school based and community interventions have not. Our project frees individuals from being alone in making subtle lifestyle changes, and uses the strength of the family unit to make changes toward healthy lifestyles. The family structure proposed in this project builds on the strengths of the family unit in Aboriginal culture, invokes role-modelling within the households and outside the household via the health counsellor, and facilitates opportunities to engage in regular group activities in a community where there is a paucity of physical activity.

This randomized controlled trial will test the feasibility of a culturally-sensitive household-based intervention, will determine the effect of the intervention on body weight, abdominal fat, blood pressure, glucose, and lipids, and will provide unique evaluation on intensive behavioural, and lifestyle modification program in a high-risk Aboriginal community.

Eligible families are randomized to intervention or control at baseline and are followed-up for 6-months. The intervention consists of: weekly home visits by trained health counsellors who provide information, advice and support on improving dietary habits and increasing physical activity; weekly home delivery of bottled water to supplant sugared drinks; and a variety of afterschool/work physical activity programs and nutritional workshops. Control families receive written material, including Canada's Food Guide to Healthy Eating and Canada's Physical Activity Guide to Healthy Active Living, which outlines suggestions for healthy living, and none of the interventions.

ELIGIBILITY:
Inclusion Criteria:

* Eligible households are defined as those comprised of a male and female parent with at least one child < 19 years old living in the same household
* Individuals between 5 and 65 years of age (including grandparents) are included
* Families must be living on Six Nations Indian Reserve, Ontario, Canada

Exclusion Criteria:

* Are not willing to have the SHARE-AP ACTION Health Counsellor visit their home on a weekly basis,
* Have a planned absence from the Reservation for > 1 month during the intervention, and
* if there is a planned break-up of the household in the next 1 year

Individual members will be excluded from the household unit if they have:

* A serious medical illness which prevent them from making dietary and exercise changes (e.g.dialysis dependent),
* Terminal cancer,
* Suspected severe alcohol abuse, or
* have suffered a recent MI or stroke in the past month.

Ages: 5 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 174
Dates: Start 2004-05; Study Completion 2005-12

PRIMARY OUTCOMES:
The primary outcomes of the pilot study include the change from baseline in daily energy intake (kcal per day), and the change in physical activity (minutes/week).

SECONDARY OUTCOMES:
Secondary outcomes include the changes (from baseline to end of study) in knowledge and attitudes toward healthy lifestyles, self/response efficacy, body fat, BMI, abdominal fat, blood pressure, glucose, and lipids.

CONTACTS AND LOCATIONS:
Overall Officials: Sonia S Anand, MD, PhD, Principal Investigator — Population Health Research Institute, McMaster University
Locations (1):
- SHARE-AP Office, Six Nations Health Services P.O. Box 5000, Ohsweken, Ontario, Canada

REFERENCES:
- [Background] Anand SS, Yusuf S, Vuksan V, Devanesen S, Teo KK, Montague PA, Kelemen L, Yi C, Lonn E, Gerstein H, Hegele RA, McQueen M. Differences in risk factors, atherosclerosis, and cardiovascular disease between ethnic groups in Canada: the Study of Health Assessment and Risk in Ethnic groups (SHARE). Lancet. 2000 Jul 22;356(9226):279-84. doi: 10.1016/s0140-6736(00)02502-2. PMID 11071182
- [Background] Davis SM, Going SB, Helitzer DL, Teufel NI, Snyder P, Gittelsohn J, Metcalfe L, Arviso V, Evans M, Smyth M, Brice R, Altaha J. Pathways: a culturally appropriate obesity-prevention program for American Indian schoolchildren. Am J Clin Nutr. 1999 Apr;69(4 Suppl):796S-802S. doi: 10.1093/ajcn/69.4.796S. PMID 10195605